CLINICAL TRIAL: NCT06614920
Title: Addressing Food-Insecurity: Plant-Based Food Prescription Program to Improve Health Food Access
Brief Title: Addressing Food Insecurity: Plant-Based Food Prescription Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: American Academy of Pediatrics (Other); Committee of Interns and Residents SEIU Healthcare (Unknown)
Responsible Party: Principal Investigator, Azaria Lewis, Internal Medicine-Pediatric Resident Physician, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20240753
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Health Literacy; Nutrition, Healthy; Nutrition Poor; Food Insecurity; Food Insecurity Among Children; Low Income Population
Keywords: Plant-based food prescription program; Plant-based; Food prescription; Food insecurity; Poverty; Nutrition education; Plant-based nutrition literacy; Plant-based nutrition education
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-Based Food Provision + Plant-Based Nutrition Education (dual intervention) (Experimental): Participants will enroll in one of four study arms based on their eligibility and interest. In Arm 1 (dual intervention- food prescription and nutrition education), we will ask participants to attend 5 nutrition classes where they will be asked to complete one survey and two brief nutrition knowledge tests (one before the class starts and one after the class is finished) each class, one survey every 3 months thereafter and one additional nutrition test 1 year after starting the program. Each class will divide participants by age (detailed in Arm 2 description).
  Participants in Arm 1 only (dual intervention) will be provided with a food prescription at the end of each class. Participants will bring this food prescription to Village FREEdge, where it will function as a voucher. Each voucher will allow for participants to pick up enough food for 6 meals per person in their household (with household maximum of 5 people)(enough meals for 3 days- 2 meals per person per day).
  Interventions: Other: Plant-Based Food Provision (with or without food prescription); Other: Plant-Based Nutrition Education
- Plant-Based Nutrition Education Only (single intervention 1) (Experimental): Participants will enroll in one of four study arms based on their eligibility and interest. In Arm 1 (dual intervention- food prescription and nutrition education) and Arm 2 (single intervention 1- nutrition education only) we will ask participants to attend 5 nutrition classes where they will be asked to complete one survey and two brief nutrition knowledge tests (one before the class starts and one after the class is finished) each class, one survey every 3 months thereafter and one additional nutrition test 1 year after starting the program. Each class will divide participants by age. If participants are 14 years old or older, they will listen to a 45-minute plant-based nutrition lecture and engage in a 45-minute interactive activity, including but not limited to plant-based meal preparation. Participants younger than 14 years old will be guided through age-appropriate interactive activities for the full 1.5-2 hours in a nearby classroom.
  Interventions: Other: Plant-Based Nutrition Education

INTERVENTIONS:
Other: Plant-Based Food Provision (with or without food prescription) — Food Prescription: Participants will bring the food prescription obtained from the nutrition class to Village FREEdge, food pantry at the Freedom Lab, where it will function as a voucher. Each voucher will allow for participants to pick up enough plant-based food for 6 meals per person in their household (with household maximum of 5 people)(enough meals for 3 days- 2 meals per person per day). We expect that participants will pick up food twice per week from Village FREEdge to obtain enough meals to feed each participant's household for 6 days out of the week for up to 1 year.
  Without food prescription: Participants will be given plant-based meals from Village FREEdge (up to two meals per day with a maximum of two meals per pick-up) without the use of a food prescription.
  Arms: Plant-Based Food Provision + Plant-Based Nutrition Education (dual intervention)
Other: Plant-Based Nutrition Education — A once weekly classes for a 5-week nutrition course. The parents/guardians would bring their children and any additional household member(s) to the nutrition class, which will organize participants in different classrooms by age (children 4 years, 4-12 years old, 12-14 years old, 14+ years old). Each classrooms will engage in age-appropriate interactive nutrition-based activities. All children below 18 will engage in interactive activities for the full 1.5 hours. Adolescents aged 14 up will join the classroom with adults and listen to a 45 minute lecture and engage in a subsequent 45 minute interactive activity that incorporates content from the lecture. The interactive activities for the children range from creating a fruit and veggie "Tik Tok" song and performing it, drawing foods on a "balanced plate", etc. The interactive activities for participants 14 year old and older range from discussions about fiber in diet, guided plant-based meal preparation, reading nutrition label etc.

SUMMARY:
Reduce food insecurity by improving plant-based health food consumption, access, health and nutrition literacy and the health of the food-insecure families we serve.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be all ages 0-99 (all arms)
* Families living under the federal poverty line AND who have food insecurity (all arms except Arm 2 which can include families with income above the federal poverty line who do not have food insecurity).
* Families cared for in either the Pediatric Mobile Clinic, Pediatric, Family Medicine, Internal Medicine or Med-Peds primary care clinics in the UHealth/Jackson Health System/Dade County Street Response.

Exclusion Criteria:

* Families who are not under the federal poverty line AND are not food insecure (all arms except Arm 2, which will include participants of all socioeconomic statuses and regardless of food security status, with no exclusion criteria in this category).
* Families who are not actively receiving outpatient primary care (all arms).

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of Servings of Unprocessed and Minimally Processed Fruits and Vegetables | Up to 1 year
  The participants will record in a weekly log the number of servings per day of unprocessed/minimally processed fruits and vegetables.
Number of Servings of Unprocessed and Minimally Processed Whole Grains | Up to 1 year
  The participants will record in a weekly log the number of servings per day of unprocessed/minimally processed whole grains.
Number of Servings of Unprocessed and Minimally Processed Legumes | Up to 1 year
  The participants will record in a weekly log the number of servings per day of unprocessed/minimally processed legumes.
Number Servings of Unprocessed and Minimally Processed Nuts/Seeds | Up to 1 year
  The participants will record in a weekly log the number of servings per day of unprocessed/minimally processed nuts/seeds.

SECONDARY OUTCOMES:
Presence of Food Insecurity | Up to 1 year
  Affirmative response to either of the two, validated screening questions for food insecurity. Investigators measured food insecurity using the validated two-question "Hunger Vital Sign" screening tool, with yes/no responses. These two questions are: "we worried whether our food would run out before we got money to buy more" and "the food we bought just didn't last and we didn't have money to get more."
Change in Plant-Based Nutrition Knowledge of Participants | Up to 1 year
  The nutrition knowledge of participants will be measured by a change in nutrition literacy pre-post test (less than 30 multiple choice questions) scores. (The pre-test will be given prior to the plant-based nutrition education course and the post-test after completion of the course).

CONTACTS AND LOCATIONS:
Overall Officials: Azaria V Lewis, DO, Principal Investigator — University of Miami
Locations (1):
- Freedom Lab 4300 NW 12th Ave, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We are not planning on sharing IPD with other researchers as that is not the arrangement of this study. We are not working with other researchers at this time.

REFERENCES:
- [Background] Bryce R, WolfsonBryce JA, CohenBryce A, Milgrom N, Garcia D, Steele A, Yaphe S, Pike D, Valbuena F, Miller-Matero LR. A pilot randomized controlled trial of a fruit and vegetable prescription program at a federally qualified health center in low income uncontrolled diabetics. Prev Med Rep. 2021 May 31;23:101410. doi: 10.1016/j.pmedr.2021.101410. eCollection 2021 Sep. PMID 34150472
- [Background] Ridberg RA, Bell JF, Merritt KE, Harris DM, Young HM, Tancredi DJ. Effect of a Fruit and Vegetable Prescription Program on Children's Fruit and Vegetable Consumption. Prev Chronic Dis. 2019 Jun 13;16:E73. doi: 10.5888/pcd16.180555. PMID 31198165
- [Background] Oronce CIA, Miake-Lye IM, Begashaw MM, Booth M, Shrank WH, Shekelle PG. Interventions to Address Food Insecurity Among Adults in Canada and the US: A Systematic Review and Meta-analysis. JAMA Health Forum. 2021 Aug 6;2(8):e212001. doi: 10.1001/jamahealthforum.2021.2001. eCollection 2021 Aug. PMID 35977189
- [Background] Bhat S, Coyle DH, Trieu K, Neal B, Mozaffarian D, Marklund M, Wu JHY. Healthy Food Prescription Programs and their Impact on Dietary Behavior and Cardiometabolic Risk Factors: A Systematic Review and Meta-Analysis. Adv Nutr. 2021 Oct 1;12(5):1944-1956. doi: 10.1093/advances/nmab039. PMID 33999108
- [Background] Xie J, Price A, Curran N, Ostbye T. The impact of a produce prescription programme on healthy food purchasing and diabetes-related health outcomes. Public Health Nutr. 2021 Aug;24(12):3945-3955. doi: 10.1017/S1368980021001828. Epub 2021 Apr 27. PMID 33902771
- [Background] Fuchs D. An overview of nutrition in medical education. JAMA. 2018;319(15):1551. doi:10.1001/jama.2018.1919.
- [Background] Centers for Disease Control and Prevention. Chronic disease prevention. Accessed January 23, 2024. Available from: https://www.cdc.gov/chronic-disease/prevention/
- [Background] Stanford Medicine. Why medical schools need to focus on nutrition. Accessed January 23, 2024. Available from: https://med.stanford.edu/school/leadership/dean/precision-health-in-the-news/why-medica-schools-need-focus-nutrition.html
- [Background] Centers for Disease Control and Prevention. Hypertension cascade: hypertension prevalence, treatment, and control estimates among US adults aged 18 years and older applying the criteria from the American College of Cardiology and American Heart Association's 2017 Hypertension Guideline-NHANES 2015-2018. US Department of Health and Human Services; 2019. Accessed January 23, 2024. Available from: https://millionhearts.hhs.gov/data-reports/hypertension-prevalence.html
- [Background] Centers for Disease Control and Prevention. Non-Hispanic Black participants had higher rates of hypertension compared to White and Hispanic participants. Accessed January 23, 2024. Available from: https://www.cdc.gov/pcd/issues/2023/23_0065.htm
- [Background] U.S. Food and Drug Administration. Improving nutrition to turn the tide on diet-related chronic disease. Accessed January 23, 2024. Available from: https://www.fda.gov/news-events/fda-voices/improving-nutrition-turn-tide-diet-related-chronic-disease
- [Background] US Burden of Disease Collaborators; Mokdad AH, Ballestros K, Echko M, Glenn S, Olsen HE, Mullany E, Lee A, Khan AR, Ahmadi A, Ferrari AJ, Kasaeian A, Werdecker A, Carter A, Zipkin B, Sartorius B, Serdar B, Sykes BL, Troeger C, Fitzmaurice C, Rehm CD, Santomauro D, Kim D, Colombara D, Schwebel DC, Tsoi D, Kolte D, Nsoesie E, Nichols E, Oren E, Charlson FJ, Patton GC, Roth GA, Hosgood HD, Whiteford HA, Kyu H, Erskine HE, Huang H, Martopullo I, Singh JA, Nachega JB, Sanabria JR, Abbas K, Ong K, Tabb K, Krohn KJ, Cornaby L, Degenhardt L, Moses M, Farvid M, Griswold M, Criqui M, Bell M, Nguyen M, Wallin M, Mirarefin M, Qorbani M, Younis M, Fullman N, Liu P, Briant P, Gona P, Havmoller R, Leung R, Kimokoti R, Bazargan-Hejazi S, Hay SI, Yadgir S, Biryukov S, Vollset SE, Alam T, Frank T, Farid T, Miller T, Vos T, Barnighausen T, Gebrehiwot TT, Yano Y, Al-Aly Z, Mehari A, Handal A, Kandel A, Anderson B, Biroscak B, Mozaffarian D, Dorsey ER, Ding EL, Park EK, Wagner G, Hu G, Chen H, Sunshine JE, Khubchandani J, Leasher J, Leung J, Salomon J, Unutzer J, Cahill L, Cooper L, Horino M, Brauer M, Breitborde N, Hotez P, Topor-Madry R, Soneji S, Stranges S, James S, Amrock S, Jayaraman S, Patel T, Akinyemiju T, Skirbekk V, Kinfu Y, Bhutta Z, Jonas JB, Murray CJL. The State of US Health, 1990-2016: Burden of Diseases, Injuries, and Risk Factors Among US States. JAMA. 2018 Apr 10;319(14):1444-1472. doi: 10.1001/jama.2018.0158. PMID 29634829